CLINICAL TRIAL: NCT00189436
Title: A Pilot Study to Evaluate the Effect of Nebulized Budesonide and Oral Corticosteroids on Wheezing Episode Relapse in Pediatric Patients Following Discharge From the Emergency Department/Outpatient Care Facility
Brief Title: Effect of Nebulized Budesonide and Oral Corticosteroids on Wheezing Episode Relapse in Children
Acronym: BudER
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Deborah Gentile (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor-Investigator, Deborah Gentile, Co-Investigator, West Penn Allegheny Health System
Organization: West Penn Allegheny Health System (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BUD ER 3425; RC - 3425 (Other: Institutional/Allegheny Singer Research Institute)
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Results first posted 2014-08-04 (Estimated); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Asthma
Keywords: Asthma
MeSH Terms: conditions — Asthma | interventions — Albuterol; Steroids

ARMS (2):
- Treatment with Budesonide (Active Comparator): Subject is treated with nebulized budesonide 0.5 BID for 3 weeks
  Interventions: Drug: Nebulized Budesonide
- Usual care (Active Comparator): Subject is treated with usual care as provided by the doctor. Usual care normally consists of treatment with albuterol with or without an oral steroid.
  Interventions: Drug: Usual care (albuterol with or without oral steroid)

INTERVENTIONS:
Drug: Nebulized Budesonide — Subject is treated with nebulized budesonide 0.5 BID for 3 weeks
  Arms: Treatment with Budesonide
Drug: Usual care (albuterol with or without oral steroid) — Subject is treated with usual care as prescribed by the doctor (normally albuterol with or without oral steroid)
  Arms: Usual care

SUMMARY:
Subjects aged 1-8 years who have been discharged from the emergency department/outpatient care facility with a diagnosis of asthma/bronchospasm/wheezing after usual standard care will be enrolled into this open-label, randomized, parallel-group study to compare the efficacy of nebulized budesonide and oral corticosteroids in preventing asthma exacerbation relapse rates during the 21-day follow-up period.

DETAILED DESCRIPTION:
Secondary outcomes include urinary cortisol-creatinine rations, symptom severity scores and peak flow rates.

ELIGIBILITY:
Inclusion Criteria:

* Children ages 1-8 years old
* Discharge from emergency department/outpatient clinic with a diagnosis of asthma exacerbation after usual standard care
* Subjects must be able to show efficient use with a jet nebulizer

Exclusion Criteria:

* Subjects requiring hospitalization
* Subjects receiving oral steroids 1 week prior to presentation to emergency department.
* Subjects with FEV1 < 50% of predicted
* Subjects with co-morbid medical conditions (renal or cardiovascular disease)
* Subjects with reported history of HIV
* Subjects unable to follow up for study visits
* Subjects who are frequently enuretic

Ages: 1 Year to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 61 (Actual)
Dates: Start 2003-03; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Skoner, MD, Principal Investigator — West Penn Allegheny Health System
Locations (2):
- United States (2):
  - Bellevue Pediatric Associates, Bellevue, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment With Budesonide | Usual Care
Started | 31 | 30
Completed | 23 | 25
Not Completed | 8 | 5

BASELINE CHARACTERISTICS:
Population: 61 subjects were enrolled and 31 were randomized to nebulized budesonide and 30 to standard of care. 74% of subjects enrolled in the nebulized budesonide and 83% enrolled in the standard care group completed the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment With Budesonide | Usual Care | Total
Number analyzed (Participants) | 31 | 30 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.8 (2.0) | 5.4 (1.6) | 5.1 (0.084)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 10 | 23
  Male | 18 | 20 | 38

OUTCOME MEASURES:

1. Primary Outcome: Wheezing/Asthma/Bronchospasm Relapse Rate
Description: This was defined as the percentage of subjects in each group (treatment with budesonide versus usual care) having an unscheduled acute visit to primary care, urgent care or an emergency department during the study period.
Time Frame: 3 weeks
Measure: Number; unit: percentage of cases of asthma relapse
Arm/Group | Treatment With Budesonide | Usual Care
Number analyzed (Participants) | 23 | 25
percentage of cases of asthma relapse | 8.7 | 4.0

2. Secondary Outcome: Urinary Cortisol Levels
Description: This was defined as the mean +/- standard deviation of 12 hour urinary cortisol levels in each group (treatment with budesonide versus usual care).
Time Frame: 3 weeks
Measure: Mean (Standard Deviation); unit: ng cortisol/mg creatinine
Arm/Group | Treatment With Budesonide | Usual Care
Number analyzed (Participants) | 23 | 25
ng cortisol/mg creatinine | 95.4 (35.3) | 141.6 (42.7)

3. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1)
Description: This was defined as the mean +/- standard deviation of FEV1 in each group (treatment with budesonide versus usual care.
Time Frame: 3 weeks
Measure: Mean (Standard Deviation); unit: % Predicted
Arm/Group | Treatment With Budesonide | Usual Care
Number analyzed (Participants) | 23 | 25
% Predicted | 86.2 (2.5) | 85.7 (3.1)

ADVERSE EVENTS:
Arm/Group | Treatment With Budesonide | Usual Care
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/30
Other Adverse Events (participants affected / at risk) | 0/31 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No